PI: Salvatore Scali

**Study Title:** Short-Term Dietary Protein Restriction Modulation of Skeletal Muscle Bioenergetics and Innate Immunity

IRB number: IRB20190098

**NCT#:** NCT03995979

<u>Statistical Analysis Plan:</u> This will be performed in a blinded fashion (no patient identifiers) by the UF Surgery Department Statistical Support Group.

## **Primary Analysis:**

Functional Enrichment Analysis using Qiagen Ingenuity Pathways Analysis; Absolute  $LogF_c$  cutoff =0.4 to describe regulation of genes; False Detection Rate (FRD)<0.1

Gene Comparison at Baseline, Day 2, Day 4, and Day 7

## Variable of Interest:

- a) Characterization of MAIT transcription response to stDR
- b) Gut microbial changes to stDR

**Additional Quantitative Analysis:** Conical Pathways and Identification of Regulators

## **Conical Pathways:**

Fischer Exact Test with FDR corrected p-value overlap threshold<0.05; Qiagen software calculations for significant pathway inhibition (negative z score) or activation (positive Z score) with |Z score|>2.0.

## **Identification of Regulators:**

Fischer Exact Test with FDR corrected p-value overlap threshold<0.01 for curated gene regulators relationships; Qiagen software calculations for significant pathway inhibition (negative z score) or activation (positive Z score) with |Z score|>2.0.